CLINICAL TRIAL: NCT02735083
Title: Long-term Follow-up Study of Patients Who Have Previously Been Exposed to UCART19 (Allogeneic Engineered T-cells Expressing a Lentiviral-based Anti-CD19 Chimeric Antigen Receptor)
Brief Title: A Study to Evaluate the Long-term Safety of Patients With Advanced Lymphoid Leukemia Who Have Been Previously Administered With UCART19
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL1-68587-003; 2016-000297-38 (EudraCT Number)
Record Dates: First submitted 2016-03-14; First posted 2016-04-12 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Advanced Lymphoid Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UCART19 follow-up (Experimental)
  Interventions: Biological: UCART19 follow-up

INTERVENTIONS:
Biological: UCART19 follow-up — UCART19 will not be administered during the study period. Patients who will be rolled-over from the parent study to this long term follow-up study, have previously received UCART19. The roll-over occurs at the end of the parent study, or at any time after UCART19 administration, in case of premature discontinuation from the parent study.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of UCART19 administration to patients with advanced lymphoid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior any study-specific procedure (patient or parent(s) or legal representative)
* Patient dosed with UCART19 who completed or discontinued early from a sponsored or from any investigator-initiated study that tested UCART19, or patients who were administered UCART19 under a special access scheme (compassionate use);
* Female patients of childbearing potential and male patients with partners of childbearing potential must continue to use an effective method of birth control as well as their partners for a 12-month duration after the last UCART19 administration.

Exclusion Criteria:

- No exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of UCART19 with or without alemtuzumab | Up to 15 Year
  * Number, duration, outcome of all adverse events (AE) within 12 months post last UCART19 infusion
  * Number, duration, outcome of adverse events of special interest (AESI) up to the end of the study
  * Proportion of patients with adverse events leading to death up to the end of the study
  * For paediatric patients: assesment of the potential impact on growth curve and puberty

SECONDARY OUTCOMES:
Assessment of long-term anti tumor activity of UCART19 | Month 3, Month 6, Month 12 during Year 1 following last UCART19 dosing then every 6 months up to Year 3, then yearly up to Year 15
Proportion of patients who underwent allogeneic HSCT (Hematopoietic Stem Cell Transplantation) for patients treated with UCART19 | Month 3, Month 6, Month 12 during Year 1 following last UCART19 dosing, then every 6 months up to Year 3, then yearly up to Year 15
Time to transplant for patients treated with UCART19 | Month 3, Month 6, Month 12 during Year 1 following last UCART19 dosing, then every 6 months up to Year 3, then yearly up to Year 15
Assessment of overall survival | Month 3, Month 6, Month 12 during Year 1 following last UCART19 dosing, then every 6 months up to Year 3, then yearly up to Year 15
Proportion of patients with detectable UCART19 levels in blood | Month 3, Month 6, Month 12 during Year 1 following last UCART19 dosing (If no more UCART19 detectable at the Month 12 visit), then every 6 months up to Year 3, then yearly up to Year 15 or the first evidence of no more detectable UCART19 (if earlier)
Proportion of patients with detectable UCART19 levels in bone marrow | Month 3, Month 6, Month 12 during Year 1 following last UCART19 dosing, then every 6 months up to Year 3, then yearly up to Year 15

CONTACTS AND LOCATIONS:
Overall Officials: Reuben Benjamin, MD, PhD, Principal Investigator — King's College Hospital NHS Trust
Locations (16):
- United States (7):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffit Cancer Center, Tampa, Florida
  - Massachussetts General Hospital, Charlestown, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (3):
  - Hôpital Saint-Louis, Paris
  - Hôpital Robert-Debré, Paris
  - Hôpital Saint-Antoine, Paris
- Japan (2):
  - Kyushyu University Hospital, Fukuoka
  - Hokkaido University Hospital, Sapporo
- Hospital San Juan De Dios, Barcelona, Spain
- United Kingdom (3):
  - King's College Hospital NHS Foundation Trust, London
  - UCL Great Ormond Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/